CLINICAL TRIAL: NCT00838812
Title: Monocentric Study, Prospective, Open and Non Controlled for to Evaluate the Effectiveness, and Tolerability the Safety of Association of Clindamycin Phosphate 1.2% and Tretinoin 0,025% in the Treatment of Acne Vulgaris Mild to Moderate, When Used Once Daily for 12 Weeks.
Brief Title: Safety and Efficacy Study of Association Between Tretinoin and Clindamycin on the Treatment of Acne Mild and Moderate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Igefarma Laboratorios S.A. (Industry)
Responsible Party: Dra. Rosa Maria Scavarelli, I
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGF 03-42008
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2010-05

CONDITIONS: Acne Vulgaris
Keywords: clindamycin; tretinoin; acne vulgaris; Acne vulgaris mild to moderate
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- clindamicin and tretinoin gel (Other)
  Interventions: Drug: application of the topic gel

INTERVENTIONS:
Drug: application of the topic gel — Clindamycin Phosphate 1,2% and tretinoin 0,025% gel once daily at night 12 weeks.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of association between tretinoin and clindamycin phosphate on the treatment of acne vulgaris mild and moderate.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes with age greater than or equal to 12 years
* Subjects diagnosed with acne vulgaris in the face, except for the nasal area, range from mild to moderate, with the following requirements.

  * Mild acne = presence of fewer than 20 comedones or less than 15 lesions, inflammatory lesions or a total of less than 30 injuries.
  * Moderate acne = presence of 20 the 100 comedones or of 15 the 50 inflamatory lesions or a total of 30 the 125 lesions, with not more than lesions small nodule until 5,0 mm.
* Ensure that the existing injuries were not submitted any treatment for acne, topical or systemic, within the last 30 days.
* Be able to properly follow the determinations of the Protocol.
* Has provided a written voluntary consent to participate in the study, by signing the informed consent, before being subjected to any procedure.
* Under 18 years old, be accompanied by legal guardian in the process of obtaining the informed consent.
* Be mentally able to provide consent and be fulfilling all the requirements of the study.

Exclusion Criteria:

* Pregnant women or in periods of lactation.
* Women of childbearing age and sexual activity with not using safe contraceptive method, such as oral contraceptives, implantable, injectable or intra-uterine, introduced for at least 120 days.
* Women who are using oral contraceptives containing the hormone combination for acetate ciprosterone and etinolestradiol, association of drospirenone and ethinyl estradiol, or desogestrel.
* Clinical evidence or history of immunodeficiency.
* Any use of immunosuppressive drug and/or immunomodulating over the past 3 months, topical or systemic.
* Concurrent use of fotossentetizadores, neuromuscular blockers, medications that exacerbate the acne, blockers (filters) with solar alcoholic vehicle, spironolactone, flutamide or zinc salts.
* Prior use of systemic retinoid.
* Presence of acne medication and/or cosmetic.
* History of systemic metabolic disorder that can interfere with the integrity of the skin.
* History of inflammatory disease, intestinal or regional enteritis and/or symptoms similar.
* History of joy to any of the components of the formula (active principle or carrier).
* History of abuse of alcohol and/or illegal drugs.
* History of non-adherence to medical treatment earlier.
* Any clinical observation made by the investigator that prohibits participation in the study of the subject.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy, through number of lesions, and tolerability of the product. | three months

CONTACTS AND LOCATIONS:
Locations (1):
- Lal Clinica, Valinhos, São Paulo, Brazil